CLINICAL TRIAL: NCT04307212
Title: Exercise is Medicine. How Exercise Signals Health Responses
Brief Title: How Exercise Signals Health Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: GFHNRC409
Record Dates: First submitted 2020-02-27; First posted 2020-03-13 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — Recombinational DNA Repair

STUDY DESIGN:
Intervention Model Description: A 3-way factorial design will be employed with training status as a between-subjects variable, and exercise intensity and time as within-subjects variables. The order of exercise intensity will be counterbalanced across subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trained (Active Comparator): Participants who have been CrossFit training at least 3 times per week for the previous 3 months. These individuals will be invited in person to participate in the study.
  Interventions: Other: 50% heart rate reserve (HRR) low intensity exercise; Other: 75% HRR moderate intensity exercise; Other: Control no exercise
- Untrained (Active Comparator): Nonactive/non--exercise trained participants who have participated in any type of exercise no more than 2 times per week for the past 3 months. These individuals will be recruited from the general public.
  Interventions: Other: 50% heart rate reserve (HRR) low intensity exercise; Other: 75% HRR moderate intensity exercise; Other: Control no exercise

INTERVENTIONS:
Other: 50% heart rate reserve (HRR) low intensity exercise — Trained and untrained participants will exercise at a constant load intensity of 50% HRR (low intensity)
Other: 75% HRR moderate intensity exercise — Trained and untrained participants will exercise at a constant load intensity of 75% HRR (moderate intensity)
Other: Control no exercise — Trained and untrained participants will have a no exercise control day

SUMMARY:
The purpose of this research is to determine the blood signals that promote health and well-being in response to exercise at different intensities.

DETAILED DESCRIPTION:
Most studies find a dose-response relationship between exercise participation and all-cause mortality. In contrast, physical inactivity and consequent overweight or obese status is associated with a cadre of health consequences. Frequently, comorbidities of obesity are mechanistically linked via chronic low grade inflammation stemming from increases in adiposity. Although exercise is known to combat obesity and obesity related disease states, the mechanisms of action are not fully understood. Therefore, the investigators propose the following study in an attempt to elucidate anti- and pro-inflammatory endocrine responses to exercise. Initial studies in animal models have provided evidence that exercise induces long-term anti-inflammatory effects, potentially via myokine signaling following skeletal muscle activation. Humans are an ideal study population as the investigators can prescribe multiple exercise protocols that mimic human behavior, and control exercise intensity to meet recommendations. Also, humans allow the investigators to collect larger plasma samples and therefore measure more circulating proteins of interest over multiple time-points. Finally, the investigators can select individuals that exercise at different frequencies, allowing the investigators to analyze the differences in endocrine responses to exercise over differing levels of fitness. In summary, a human model will allow for a much better understanding of the human condition.

ELIGIBILITY:
Inclusion Criteria:

* No tobacco use
* Not pregnant, lactating, or planning to become pregnant in the next 6 months
* Regular menses for the past 6 months
* No use of hormone replacement for metabolic conditions (use of hormonal contraceptives are not exclusionary)
* No physical limitations
* Has the ability to safely perform exercise

Exclusion Criteria:

* Has no major health problems
* Cannot have known cardiovascular (cardiac, peripheral vascular, cerebrovascular), pulmonary (COPD, interstitial lung disease, cystic fibrosis) or metabolic (diabetes, thyroid disorders, renal or liver disease) disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Change in plasma myokine concentration | Pre-exercise, 0, 30, 60, 90 minutes post-exercise
  Blood samples collected during exercise will be analyzed for the concentration of plasma myokines including Brain Derived Neurotropic Factor (BDNF), Secreted Protein Acidic and Rich in Cysteine (SPARC), Leukemia Inhibitory Factor (LIF), Interleukin (IL) 15, IL-6, Myostatin, Irisin, Follistatin-like 1 (FSTL-1), Fibroblast Growth Factor 21 (FGF-21), IL-4, IL-7 receptor agonist (ra), IL-7, beta-aminoisobutyric acid (BAIBA), IL-1ra, Growth Differentiation Factor (GDF) 8, Insulin-Like Growth Factor-1 (IGF1).

SECONDARY OUTCOMES:
Change in plasma adipokine concentration | Pre-exercise, 0, 30, 60, 90 minutes post-exercise
  Blood samples collected during exercise will be analyzed for the concentration of plasma adipokines including myonectin.
Change in plasma cytokine concentration | Pre-exercise, 0, 30, 60, 90 minutes post-exercise
  Blood samples collected during exercise will be analyzed for the concentration of plasma cytokines including IL-8, Tumor necrosis factor alpha (TNFα), C-reactive protein (CRP), fibrinogen, and IGF1.
Relative reinforcing value (RRV) of exercise | Week 0
  RRV of exercise will be assessed by evaluating the number of responses (mouse button presses) a participant is willing to complete to gain access to exercise or an alternative (magazines, word games, puzzles).
Minutes of physical activity, as assessed by activity tracker | Week 0
  Minutes of physical activity will be assessed by having participants wear an Actigraph accelerometer for 7 days (minimum 10 hours per day) on the right hip.
Usual modes of sedentary behavior | Week 0
  Usual modes of sedentary behavior will be determined via the validated International Physical Activity Questionnaire (IPAQ). The IPAQ measures habitual physical activity for the past 7 days and consists of four domains of physical activity: job-related (7 items), transportation (6 items), household/gardening (6 items), and leisure-time activities (6 items). To show sedentary behavior, two questions regarding time spent sitting are also included. The number of minutes for each activity class is multiplied by the MET score for that activity to convert the IPAQ data into metabolic equivalent scores (MET-min-week-1). Physical activity levels are then classified as being inactive, minimally active, and health-enhancing physically active.
Preference for intense physical activity and tolerance for exercise discomfort | Week 0
  Preference for intense physical activity and tolerance for exercise discomfort will be assessed by self-report questionnaire responses to the Preference for and Tolerance of the Intensity of Exercise Questionnaire (PRETIE-Q). The PRETIE-Q measures preference for high intensity vs. low intensity exercise and ability to persist or tolerate the discomfort associated with intense exercise. The PRETIE-Q consists of two subscales: Preference for Exercise Intensity and Tolerance of Exercise Intensity. Each subscale has 8 items rated on a 5-point response scale (range 8 - 40). Higher scores indicate greater preference for intense exercise and/or greater tolerance for exercise discomfort. Total scale scores are not used. Scale averages will be used.
Fat mass as assessed by dual energy x-ray absorptiometry (DXA) scans | Week 0
  Participants will be instructed to lie supine with hands by their sides on a GE Lunar iDXA machine for a full-body x-ray scan which will measure grams and percentage changed in fat mass.
Fat-free lean mass as assessed by DXA scans | Week 0
  Participants will be instructed to lie supine with hands by their sides on a GE Lunar iDXA machine for a full-body x-ray scan which will measure grams and percentage changed in fat-free lean mass.

CONTACTS AND LOCATIONS:
Overall Officials: James Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: USDA Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT04307212/ICF_000.pdf